CLINICAL TRIAL: NCT05224479
Title: Clinical Validation of Machine Learning Triage of Chest Radiographs
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in research plan
Sponsor: Stanford University (Other)
Collaborators: Society of Thoracic Radiology (Unknown)
Responsible Party: Principal Investigator, Emily Tsai, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 47832
Record Dates: First submitted 2022-01-22; First posted 2022-02-04 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Chest--Diseases

STUDY DESIGN:
Intervention Model Description: Radiologists will triage chest radiographs using traditional, machine learning, and random methods.
Who Masked: Participant
Masking Description: Radiologists will be blinded when using machine learning and random triage methods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional workflow triage (Active Comparator): Radiologists follow standard triage of chest radiographs.
  Interventions: Other: Traditional workflow triage; Other: Machine learning workflow triage; Other: Random workflow triage
- Machine learning workflow triage (Active Comparator): Radiologists follow machine learning triage of chest radiographs.
  Interventions: Other: Traditional workflow triage; Other: Machine learning workflow triage; Other: Random workflow triage
- Random workflow triage (Sham Comparator): Radiologists follow randomly ordered triage of chest radiographs.
  Interventions: Other: Traditional workflow triage; Other: Machine learning workflow triage; Other: Random workflow triage

INTERVENTIONS:
Other: Traditional workflow triage — Workflow triage is based on order location, STAT designation, and first-in-first-out status.
Other: Machine learning workflow triage — Workflow triage is based on the machine learning model's confidence of abnormality.
Other: Random workflow triage — Workflow triage is based on random order.

SUMMARY:
Artificial intelligence and machine learning have the potential to transform the practice of radiology, but real-world application of machine learning algorithms in clinical settings has been limited. An area in which machine learning could be applied to radiology is through the prioritization of unread studies in a radiologist's worklist. This project proposes a framework for integration and clinical validation of a machine learning algorithm that can accurately distinguish between normal and abnormal chest radiographs. Machine learning triage will be compared with traditional methods of study triage in a prospective controlled clinical trial. The investigators hypothesize that machine learning classification and prioritization of studies will result in quicker interpretation of abnormal studies. This has the potential to reduce time to initiation of appropriate clinical management in patients with critical findings. This project aims to provide a thoughtful and reproducible framework for bringing machine learning into clinical practice, potentially benefiting other areas of radiology and medicine more broadly.

ELIGIBILITY:
Inclusion Criteria:

* Radiologist at Stanford Hospital and Clinics

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Turnaround time | up to 1 hour
  Time from completion of radiograph to time that radiologist issues an assessment via preliminary or final report

CONTACTS AND LOCATIONS:
Overall Officials: Emily Tsai, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No